CLINICAL TRIAL: NCT01532167
Title: Impact and Utility of Positron Emission Tomography (PET) for the Assessment of Inflammatory Activity Arteritis Versus Clinical Score and Laboratory Values in Takayasu Arteritis: a Cohort Study
Brief Title: Impact and Utility of PET Versus Clinical Score for the Assessment of Inflammatory Activity in Takayasu Arteritis
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Jose Telich, Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 12-755
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate that [18F]FDG PET is a a better method than clinical and laboratory values for the identification and assessment of inflammatory activity in patients with Takayasu Arteritis (TA), allowing long-term follow-up with a precise evaluation of response to therapy.

DETAILED DESCRIPTION:
Inflammatory activity and fibrosis are the main causes of morbidity and mortality in patients with Takayasu arteritis. The investigators objective is to determine the utility of using 18F-FDG PET in the basal evaluation and follow-up of patients and compare the results with Dabague's clinical score.

ELIGIBILITY:
Inclusion Criteria:

* TA was diagnosed if the patient met 3 or more ACR criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for TA at our institution's immunology outpatient clinic were included between.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Soto, MD, Principal Investigator — Instituto Nacional de Cardiologia; Erick Alexanderson, MD, Study Director — Instituto Nacional de Cardiologia
Locations (1):
- Instituto Nacional de Cardiologia, Mexico City, Mexico City, Mexico